CLINICAL TRIAL: NCT02629718
Title: A Trial of Neoadjuvant Chemotherapy Followed by Surgery Versus Surgery in FIGO IB2 and IIA2 Cervical Cancer(CSEM005)
Brief Title: Neoadjuvant Chemotherapy + Surgery Versus Surgery in FIGO IB2 and IIA2 Cervical Cancer
Acronym: SYSGO-003
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-FXY-069
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: PFS; OS; Quality of Life
Keywords: neoadjuvant chemotherapy; radical surgery; cervical carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(NACT) (Experimental): Neoadjuvant Chemotherapy followed by Radical Surgery
  Interventions: Drug: NACT (Paclitaxel + Cisplatin or carboplatin); Procedure: radical surgery
- B(RS) (Active Comparator): Radical Surgery alone
  Interventions: Procedure: radical surgery

INTERVENTIONS:
Drug: NACT (Paclitaxel + Cisplatin or carboplatin) — Paclitaxel 150mg/m2 over 3 hours + Cisplatin 70mg/m2 or carboplatin AUC = 6, repeat per 21 days, 3 cycles.
  Arms: A(NACT)
Procedure: radical surgery — Radical hysterectomy (Piver Type III or Type IV hysterectomy) plus bilateral pelvic lymph node dissection and para-aortic lymph node dissection or sampling

SUMMARY:
To clarify the potential benefits of NACT before radical surgery(RS), we perform a phase III, randomised controlled trial to compare NACT plus RS with RS alone in patients with stages IB2 and IIA2 cervical cancer.

DETAILED DESCRIPTION:
Patients with International Federation of Gynecology and Obstetrics (FIGO) stage IB2 and IIA2 cervical cancer are eligible for our study. They will receive paclitaxel + cisplatin(TP)/carboplatin(TC) regimen neoadjuvant chemotherapy (NACT) 3 cycles followed by radical surgery (RS) (type III to V radical hysterectomy plus systematic pelvic lymphadenectomy) (arm A) or directly radical surgery (arm B). Postoperative pelvic radiotherapy will be started within 6 weeks after surgery if the patients have pelvic lymph node metastasis, parametrial involvement, deep stromal invasion or positive margin. Extended-field external beam therapy, delivering a dose of 4500cGy by a four-field technique, will be administered to patients with positive para-aortic nodes. High-dose rate brachytherapy will be delivered to the vaginal stump if patients have positive surgical margins. The primary end point is 2-years progression-free survival, The secondary end points is overall survival , rate of response to TP or TC regimen chemotherapy and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed cervical carcinoma;
* Histopathology squamaous carcinoma, adenocarcinoma or adeno-squamous carcinoma;
* Original clinical stage must be IB2 or IIA2 （FIGO);
* Age between 18-65;
* Patients must give signed informed consent;
* P.S status: 0-1;
* Estimated survival time > 3 months;

Exclusion Criteria:

* The presence of uncontrolled life-threatening illness;
* Receiving other ways of anti-cancer therapy;
* Investigator consider the patients can't finish the whole study;
* With normal liver function test (ALT、AST>2.5×ULN);
* With normal renal function test (Creatinine>1.5×ULN);
* WBC<4,000/mm3 or PLT<100,000/mm;
* Accompany with other malignancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2015-12; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 years

SECONDARY OUTCOMES:
overall survival | 5 years
quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Department of Gynecologic Oncology, Guangzhou, Guangdong, China